CLINICAL TRIAL: NCT01288716
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Tolerability of STX209 (Arbaclofen) Administered for the Treatment of Social Withdrawal in Subjects With Autism Spectrum Disorders
Brief Title: Study of Arbaclofen for the Treatment of Social Withdrawal in Subjects With Autism Spectrum Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seaside Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 209AS208
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Autism Spectrum Disorders
Keywords: ASD; Autism; Asperger Syndrome
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome | interventions — arbaclofen placarbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
- Arbaclofen (Active Comparator)
  Interventions: Drug: Arbaclofen

INTERVENTIONS:
Drug: Arbaclofen
  Other Names: STX209, R-baclofen
  Arms: Arbaclofen

SUMMARY:
To explore the efficacy, safety and tolerability of STX209 (arbaclofen) administered for the treatment of social withdrawal in subjects with autism spectrum disorders

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorders (ASD)
* Current pharmacological treatment regimen has been stable for at least 4 weeks prior to Screening.
* Subjects with a history of seizure disorder must currently be receiving treatment with antiepileptics and must have been seizure free for 6 months, or must be seizure free for 3 years if not currently receiving antiepileptics.
* If the subject is already receiving stable non-pharmacologic educational, behavioral, and/or dietary interventions, participation in these programs must have been continuous during the 2 months prior to Screening

Exclusion Criteria:

* Subjects with any condition, including alcohol and drug abuse, which might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being.
* Subjects who plan to initiate or change pharmacologic or non-pharmacologic interventions during the course of the study.
* Subjects who have taken another investigational drug within the last 30 days.
* Subjects who are not able to take oral medications

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist-Social Withdrawal Subscale | At 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - University of California-Los Angeles Neuropsychiatric Institute, Los Angeles, California
  - University of California-Davis, M.I.N.D. Institute, Sacramento, California
  - Pharmax Research Clinic, Miami, Florida
  - Lake Mary Pediatrics, Orange City, Florida
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - Institute for Juvenile Research, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Missouri, Thompson Research Center for Autism & Neurodevelpmental Disorders, Columbia, Missouri
  - Seaver Autism Center, Mount Sinai Medical Center, New York, New York
  - University of North Carolina Neurosciences Hospital, Chapel Hill, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cutting Edge Research, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Tennessee Medical Group, LeBonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt Kennedy Center, Nashville, Tennessee
  - Red Oaks Psychiatry Associates, P.A., Houston, Texas
  - Road Runner Research, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington